CLINICAL TRIAL: NCT00167700
Title: Nutrition, Allergy, Mucosal Immunology and Intestinal Microbiota (NAMI): Pre-, Peri- and Postnatal Programming and Origins of Disease: Early Targeting the Epidemics of Allergy and Overweight
Brief Title: Pre-, Peri- and Postnatal Programming and Origins of Disease: Early Targeting the Epidemics of Allergy and Overweight
Acronym: NAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15214
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Disease; Obesity; Immunology
Keywords: atopic disease; probiotics; gut microbiota; allergy; nutrition; growth; allergic rhinitis; atopic sensitization; risk-markers of life-style related diseases
MeSH Terms: conditions — Obesity; Hypersensitivity; Rhinitis, Allergic | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Probiotics (Experimental)
  Interventions: Dietary Supplement: Probiotics
- Probiotics + Dietary counseling (Experimental)
  Interventions: Behavioral: Dietary counselling and probiotics
- Dietary counseling + placebo (Experimental)
  Interventions: Behavioral: Dietary counselling and placebo
- Prebiotics (Experimental)
  Interventions: Dietary Supplement: Prebiotics
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo capsules
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Dietary counselling and placebo — Counseling to conform with the dietary recommendations. Food products commercially available including spreads and salad dressing. Placebo capsules.
  Arms: Dietary counseling + placebo
Behavioral: Dietary counselling and probiotics — Counseling to conform with the dietary recommendations. Food products commercially available including spreads and salad dressing. Probiotics
  Arms: Probiotics + Dietary counseling
Dietary Supplement: Placebo capsules — Placebo capsules
  Arms: Placebo
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Prebiotics
  Arms: Prebiotics

SUMMARY:
Combined programme: Nutrition, Allergy, Mucosal immunology and Intestinal microbiota (NAMI) was created with the objective to reverse the rising trend of chronic inflammatory diseases, such as allergic disease and obesity, by control of the internal and external environments of the infant. To approach this problem, the project aims to characterize

* how immunology is regulated during pregnancy and early infancy,
* how the immune interaction between mother and child is influenced by nutritional and microbial factors, and
* how the regulation is related to disease risk.

DETAILED DESCRIPTION:
While allergic diseases comprise the most common chronic disease in childhood, obesity is the most prevalent nutritional disorder among children throughout the world. In Europe, an estimated 20% of children and adolescents are overweight with one-third of these being considered obese. Moreover, escalation of these problems is expected in the future, since the velocity of propagation is highest in children. Although genetic factors can determine the propensity of an individual to become allergic or obese, these unlikely explain the recent and progressive worldwide increases in incidence. Rather, it would appear that the environmental changes more directly shape the risk during a critical period of life when the scene is set for the consolidation of the immune responder type. Prenatal environmental exposures may alter gene expression via epigenetic mechanisms, heritable changes in gene expression occurring without alterations in the DNA sequences.

Specifically current research interest is directed towards health promotion and reducing the risk of disease evaluating the probiotic effects with specific foods and nutrients, and assessing their interactions in optimal combination and food matrix. For this purpose a series of interventions studies evaluate the both the optimal timing of probiotic intervention and the optimal mode of administration.

Sections:

Prenatal

RCT 2 Randomized, parallel-design clinical trial of 3 groups. Pregnant women (n=256) from families with at least one member having an allergic disease have been recruited from maternal welfare clinics and randomly assigned to control group or one of the intervention groups. Mothers in the dietary intervention groups received dietary counselling with specific attention to the quality and quantity of fat in the diet. To promote the achievement of current dietary recommendations, mothers have been provided with foods which have a favourable fat composition (e.g. spreads). The subjects in the intervention groups have been further randomized (double-blind randomization) to receive either placebo or a probiotic preparation, 1010 cfu of both Lactobacillus rhamnosus GG and Bifidobacterium lactis and controls received placebo in a single-blind manner. Dietary food products and probiotic supplementation have been continued from the 1st trimester of pregnancy until the end of exclusive breast feeding, maximum of 6 months.

Perinatal

RCT 1 Randomized double-blind, placebo-controlled study of 2 groups. Pregnant women (n=159) have been randomized into one of the study groups 2-4 weeks before term to receive placebo (microcrystalline cellulose) or probiotic Lactobacillus rhamnosus GG (ATCC 53103; 1010 cfu). After delivery probiotics/ placebo were administered orally to the infants for 6 months. General information to prevent allergy has been given in written form to all: to breast-feed for at least 4-6 months; to begin solid foods at 4-6 months; no smoking by caretakers.

RCT 3 Randomized double-blind, placebo-controlled clinical trial of 3 groups. Pregnant women (n=241) with a history of atopic diseases have been assigned to one of the treatment groups: to receive for 2 months before delivery and for 2 months thereafter, when they are breast-feeding, either placebo or Lactobacillus rhamnosus and Bifidobacterium longum or Lactobacillus paracasei and Bifidobacterium longum.

Postnatal

RCT 4 Randomized double-blind, placebo-controlled study of 3 groups. Neonates (n=94) fulfilling the following criteria: gestational age at birth between 32nd and 36th weeks, weight over 1500 g and no congenital defects of gastrointestinal system or other defects that prevent enteral nutrition, have been randomized to receive either placebo (microcrystalline cellulose) or a probiotic preparation (Lactobacillus rhamnosus GG, ATCC 53103) or a prebiotic preparation (a mixture of Polydextrose and Galacto-oligosaccharideOS in a 1:1 ratio). The treatment continues for 2 months.

RCT 5 Randomized double-blind, placebo-controlled clinical trial of 2 groups. 2-6 weeks old formula- and breast-fed colic infants (n=30), who cry without medical cause for 3h/d, for 3days/week, have been randomized to receive either placebo (microcrystalline cellulose) or a probiotic preparation (Lactobacillus rhamnosus GG, ATCC 53103) for 4 weeks. Formula-fed infants receive extensively hydrolysed formula and mothers of breast-fed infants avoid cow's milk in their diet.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from families with at least one family member having an allergic disease

Exclusion Criteria:

* Women presenting severe immunological or other chronic diseases (rheumatoid arthritis, diabetes, inflammatory bowel disease, thyroid diseases, malignancies etc.)
* Women who cannot be expected to comply with treatment
* Women currently participating or having participated in other clinical trial during the last 2 months prior to the beginning of the intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1997-02; Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with allergic disease | Up to 13 years
Weight gain | Up to 13 years
Number of patients with chronic inflammatory disease | Up to 13 years

SECONDARY OUTCOMES:
Innate immune gene expression patterns | Up to 13 years
Microbiota composition
  Amount of bacterial cells (per gram of faeces of mothers and infants as well as of breast milk) is measured using multiple methods, i.e. pyrosequencing, HIT-CHIP, qPCR, FISH and DGGE.
Plasma glucose | Up to 13 years
Cytokines in peripheral blood | Up to 13 years
Cytokine profile in breast milk | Up to 13 years
Cytokine profile in peripheral blood mononuclear cells (PBMC) | Up to 13 years
GHbA1c | Up to 13 years
Fatty acids | Up to 13 years
Lipoproteins | Up to 13 years
Intakes of foods and nutrients | Up to 13 years
Blood pressure | Up to 13 years
Leukotrienes in peripheral blood | Up to 13 years
Adipokines | Up to 13 years
Amount of crying in minutes | Up to 1 year
  Crying minutes per day
Number of patients with functional gastrointestinal disorders | Up to 13 years
Incidence of viral infections | Up to 13 years

CONTACTS AND LOCATIONS:
Overall Officials: Erika Isolauri, MD, PhD, Study Director — University of Turku
Locations (1):
- Turku University Central Hospital, Turku, Finland

REFERENCES:
- [Result] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Result] Kalliomaki M, Salminen S, Poussa T, Arvilommi H, Isolauri E. Probiotics and prevention of atopic disease: 4-year follow-up of a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1869-71. doi: 10.1016/S0140-6736(03)13490-3. PMID 12788576
- [Result] Laiho K, Lampi AM, Hamalainen M, Moilanen E, Piironen V, Arvola T, Syrjanen S, Isolauri E. Breast milk fatty acids, eicosanoids, and cytokines in mothers with and without allergic disease. Pediatr Res. 2003 Apr;53(4):642-7. doi: 10.1203/01.PDR.0000055778.58807.C8. Epub 2003 Jan 29. PMID 12612204
- [Result] Laitinen K, Kalliomaki M, Poussa T, Lagstrom H, Isolauri E. Evaluation of diet and growth in children with and without atopic eczema: follow-up study from birth to 4 years. Br J Nutr. 2005 Oct;94(4):565-74. doi: 10.1079/bjn20051503. PMID 16197582
- [Result] Collado MC, Laitinen K, Salminen S, Isolauri E. Maternal weight and excessive weight gain during pregnancy modify the immunomodulatory potential of breast milk. Pediatr Res. 2012 Jul;72(1):77-85. doi: 10.1038/pr.2012.42. Epub 2012 Mar 27. PMID 22453296
- [Result] Laitinen K, Poussa T, Isolauri E; Nutrition, Allergy, Mucosal Immunology and Intestinal Microbiota Group. Probiotics and dietary counselling contribute to glucose regulation during and after pregnancy: a randomised controlled trial. Br J Nutr. 2009 Jun;101(11):1679-87. doi: 10.1017/S0007114508111461. Epub 2008 Nov 19. PMID 19017418
- [Result] Hoppu U, Isolauri E, Laakso P, Matomaki J, Laitinen K. Probiotics and dietary counselling targeting maternal dietary fat intake modifies breast milk fatty acids and cytokines. Eur J Nutr. 2012 Mar;51(2):211-9. doi: 10.1007/s00394-011-0209-0. Epub 2011 May 31. PMID 21626296
- [Result] Niinivirta K, Isolauri E, Laakso P, Linderborg K, Laitinen K. Dietary counseling to improve fat quality during pregnancy alters maternal fat intake and infant essential fatty acid status. J Nutr. 2011 Jul;141(7):1281-5. doi: 10.3945/jn.110.137083. Epub 2011 May 18. PMID 21593355
- [Result] Ilmonen J, Isolauri E, Poussa T, Laitinen K. Impact of dietary counselling and probiotic intervention on maternal anthropometric measurements during and after pregnancy: a randomized placebo-controlled trial. Clin Nutr. 2011 Apr;30(2):156-64. doi: 10.1016/j.clnu.2010.09.009. PMID 20970896
- [Result] Luoto R, Laitinen K, Nermes M, Isolauri E. Impact of maternal probiotic-supplemented dietary counseling during pregnancy on colostrum adiponectin concentration: a prospective, randomized, placebo-controlled study. Early Hum Dev. 2012 Jun;88(6):339-44. doi: 10.1016/j.earlhumdev.2011.09.006. Epub 2011 Sep 25. PMID 21945174
- [Result] Ojala T, Aaltonen J, Siira S, Jalonen J, Ekholm E, Ekblad U, Laitinen K. Fetal cardiac sympathetic activation is linked with maternal body mass index. Early Hum Dev. 2009 Sep;85(9):557-60. doi: 10.1016/j.earlhumdev.2009.05.009. Epub 2009 Jun 12. PMID 19524376
- [Result] Luoto R, Laitinen K, Nermes M, Isolauri E. Impact of maternal probiotic-supplemented dietary counselling on pregnancy outcome and prenatal and postnatal growth: a double-blind, placebo-controlled study. Br J Nutr. 2010 Jun;103(12):1792-9. doi: 10.1017/S0007114509993898. Epub 2010 Feb 4. PMID 20128938
- [Result] Collado MC, Isolauri E, Laitinen K, Salminen S. Effect of mother's weight on infant's microbiota acquisition, composition, and activity during early infancy: a prospective follow-up study initiated in early pregnancy. Am J Clin Nutr. 2010 Nov;92(5):1023-30. doi: 10.3945/ajcn.2010.29877. Epub 2010 Sep 15. PMID 20844065
- [Result] Aaltonen J, Ojala T, Laitinen K, Poussa T, Ozanne S, Isolauri E. Impact of maternal diet during pregnancy and breastfeeding on infant metabolic programming: a prospective randomized controlled study. Eur J Clin Nutr. 2011 Jan;65(1):10-9. doi: 10.1038/ejcn.2010.225. Epub 2010 Oct 13. PMID 20948557
- [Derived] Luoto R, Partty A, Vogt JK, Rautava S, Isolauri E. Reversible aberrancies in gut microbiome of moderate and late preterm infants: results from a randomized, controlled trial. Gut Microbes. 2023 Dec;15(2):2283913. doi: 10.1080/19490976.2023.2283913. Epub 2023 Nov 27. PMID 38010080
- [Derived] Davidson SJ, Barrett HL, Price SA, Callaway LK, Dekker Nitert M. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD009951. doi: 10.1002/14651858.CD009951.pub3. PMID 33870484
- [Derived] Partty A, Kalliomaki M, Salminen S, Isolauri E. Infantile Colic Is Associated With Low-grade Systemic Inflammation. J Pediatr Gastroenterol Nutr. 2017 May;64(5):691-695. doi: 10.1097/MPG.0000000000001340. PMID 27478897
- [Derived] Partty A, Lehtonen L, Kalliomaki M, Salminen S, Isolauri E. Probiotic Lactobacillus rhamnosus GG therapy and microbiological programming in infantile colic: a randomized, controlled trial. Pediatr Res. 2015 Oct;78(4):470-5. doi: 10.1038/pr.2015.127. Epub 2015 Jul 7. PMID 26151493
- [Derived] Luoto R, Ruuskanen O, Waris M, Kalliomaki M, Salminen S, Isolauri E. Prebiotic and probiotic supplementation prevents rhinovirus infections in preterm infants: a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2014 Feb;133(2):405-13. doi: 10.1016/j.jaci.2013.08.020. Epub 2013 Oct 13. PMID 24131826
- [Derived] Partty A, Luoto R, Kalliomaki M, Salminen S, Isolauri E. Effects of early prebiotic and probiotic supplementation on development of gut microbiota and fussing and crying in preterm infants: a randomized, double-blind, placebo-controlled trial. J Pediatr. 2013 Nov;163(5):1272-7.e1-2. doi: 10.1016/j.jpeds.2013.05.035. Epub 2013 Jul 31. PMID 23915796
- [Derived] Cabrera-Rubio R, Collado MC, Laitinen K, Salminen S, Isolauri E, Mira A. The human milk microbiome changes over lactation and is shaped by maternal weight and mode of delivery. Am J Clin Nutr. 2012 Sep;96(3):544-51. doi: 10.3945/ajcn.112.037382. Epub 2012 Jul 25. PMID 22836031
- [Derived] Grzeskowiak L, Collado MC, Mangani C, Maleta K, Laitinen K, Ashorn P, Isolauri E, Salminen S. Distinct gut microbiota in southeastern African and northern European infants. J Pediatr Gastroenterol Nutr. 2012 Jun;54(6):812-6. doi: 10.1097/MPG.0b013e318249039c. PMID 22228076
- [Derived] Grzeskowiak L, Gronlund MM, Beckmann C, Salminen S, von Berg A, Isolauri E. The impact of perinatal probiotic intervention on gut microbiota: double-blind placebo-controlled trials in Finland and Germany. Anaerobe. 2012 Feb;18(1):7-13. doi: 10.1016/j.anaerobe.2011.09.006. Epub 2011 Sep 29. PMID 21979491
- [Derived] Huurre A, Kalliomaki M, Rautava S, Rinne M, Salminen S, Isolauri E. Mode of delivery - effects on gut microbiota and humoral immunity. Neonatology. 2008;93(4):236-40. doi: 10.1159/000111102. Epub 2007 Nov 16. PMID 18025796